CLINICAL TRIAL: NCT04054180
Title: Multimodal Remote Monitoring and Integrated Educational Program in OSA Patients Initiating Continuous Positive Airway Pressure (CPAP): a Prospective Intervention (SLEEPCONNECT)
Brief Title: Multimodal Remote Monitoring and Integrated Educational Program in OSA Patients Initiating Continuous Positive Airway Pressure (CPAP): (SLEEPCONNECT)
Acronym: SLEEPCONNECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Grenoble (Other)
Collaborators: SEFAM MEDICAL (Villiers les Nancy, France) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC18.338
Record Dates: First submitted 2019-07-29; First posted 2019-08-13 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Continuous positive airway pressure; Connected devices
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Weights and Measures; Fitness Trackers

STUDY DESIGN:
Intervention Model Description: This is a prospective, open, multicentric, national and uncontrolled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP S.Box associated with its 3 connected devices (Experimental): S.BOXTM CPAP associated with its 3 connected devices Each patient will be monitored by a CPAP S.Box, with a Sefam Access application installed on their Smartphone to collect data from 3 connected measuring devices: PROMs, an activity monitor and a blood pressure monitor.
  Interventions: Other: CPAP associated with connected devices: blood pressure monitor , scales and activity monitor

INTERVENTIONS:
Other: CPAP associated with connected devices: blood pressure monitor , scales and activity monitor — CPAP associated with connected devices: blood pressure monitor , PROMs and activity monitor Patients will use their connected devices for one year. Data from the connected devices will be transmitted to their smartphone application Sefam Access. At the beginning of the study, patients will have a dietary assessment and start a support program for nutrition counselling and physical activity. At each study visit the dietician and physical exercise coach will give the patient advices on diet and for adjusting physical activity.

SUMMARY:
Continuous positive airway pressure (CPAP) is the first line therapy for Obstructive Sleep Apnea Syndrome (OSAS) but has limited impact for reducing cardio-metabolic risk.

Combined treatment strategies including physical activity and weight loss management have emerged in association with CPAP. Patient's engagement might be supported by connected devices and smartphone applications measuring physical activity, blood pressure, weight and sleep duration. Data fusion of these parameters with CPAP-remote telemonitoring will allow personalized coaching and integrated care of OSAS with cardio-metabolic co-morbidities.

DETAILED DESCRIPTION:
"SLEEPCONNECT" is a prospective multicenter observational study with:

* Evaluation of the impact of multimodal remote monitoring using connected devices and a dedicated smartphone application on the control of blood pressure after 3 months of CPAP.
* Evaluation of impact of such an integrated care on physical activity and body weight

This study is supported by the S.BOXTM CPAP device and its companion connected devices (physical activity, blood pressure, sleep duration, weight) and smartphone application collecting CPAP telemonitoring and assessing patients reported outcomes (PROMs). Patients have a continuous access to their own data.

Digital health system will be complemented by physical activity and nutrition coaching. Coaching persons will be inform during the follow-up by data collected by connected devices and app.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea syndrome not treated with CPAP and defined by an apnea-hypopnea index (AHI) greater than 15 events per hour and with more than 80% of obstructive events, determined by polysomnography (PSG) or polygraphy (PG) within the last 6 months
* Treated hypertension or newly diagnosed hypertension defined as 140 ≤ SBP <180 mmHg and 90 ≤ DBP<110 mmHg
* BMI > 28 kg / m²
* Smartphone
* Able to use a mobile application on a personal smartphone
* Medical certificate for the practice of physical activity/exercise
* Patients who have freely given their informed written consent
* Person affiliated to the French social security system

Exclusion Criteria:

* Central sleep apnea syndrome
* Patient with planned bariatric surgery
* Severe bullous emphysema
* Pneumothorax
* Trauma or recent surgery to or affecting the forebrain with sequelae of cranio-naso/pharyngeal fistula
* Decompensated cardiac insufficiency or hypotension, particularly in the event of reduced blood volume or in the case of cardiac arrhythmias
* Dehydration
* Tracheotomy
* Pregnant or lactating women
* Patient currently participating or having participated in the month prior to inclusion in another interventional clinical research project that may impact the study
* Patients under guardianship or curatorship
* Patients not affiliated to the French social security system or equivalent
* Patients deprived of their liberty or hospitalized without their consent
* Major patients protected by law
* Person under administrative or judicial review
* Minor patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of mean value of 18 self measures blood pressure | baseline and 3 months
  Patients will have a connected blood pressure monitor and will make self-measurements at inclusion and 3 months after starting CPAP.
  Self-measurement consists of 3 measurements, with a 1 minute interval between each one, each morning and evening over 3 days.

SECONDARY OUTCOMES:
Comparison of variability of 18 measurements of SBP by self-measurement, between inclusion and after 3 months of CPAP treatment | baseline to 3 months
  Patients will have a connected blood pressure monitor and will be asked to make self-measurements at baseline and at 15 days, 1 month, 2 months, and 3 months after starting CPAP.
Comparison of variability of 18 measurements of DBP by self-measurement, between inclusion and after 3 months of CPAP treatment | baseline to 3 months
  Patients will have a connected blood pressure monitor and will be asked to make self-measurements at baseline and at 15 days, 1 month, 2 months, and 3 months after starting CPAP.
Comparison of variability of 18 measurements of mean blood pressure by self-measurement, between inclusion and after 3 months of CPAP treatment | baseline to 3 months
  Patients will have a connected blood pressure monitor and will be asked to make self-measurements at baseline and at 15 days, 1 month, 2 months, and 3 months after starting CPAP.
Comparison of number of steps measured before initiating CPAP and at 3 months | baseline and 3 months
  Patients will be required to wear their connected activity monitor for one week at inclusion, and 3 months of CPAP treatment.
Evaluation of change in biological laboratory parameters | baseline and 3 months
  Comparison of fasting glucose between baseline and after 3 months of CPAP treatment
Evaluation of change in biological laboratory parameters | baseline and 3 months
  Comparison of lipid profile between baseline and after 3 months of CPAP treatment
Weight variation over three months | baseline and 3 months
  Weight will be recorded using their connected devices at baseline, and 3 months of CPAP treatment.
Assessment of reasons for refusal of digital health by a dedicated questionnaire conducted in patients who refused to participate in the study | baseline
  Thirteen questions about: sex, age, professional status, employment situation, smartphone usages, frequency of smartphone use, connected devices and opinions on this.
Comparison of residual AHI between Polylink respiratory polygraphic data and AHI measurement by CPAP S.Box | 24 hours
  After 3 months of treatment by CPAP the patient will have a home polygraphy using the Polylink polygraph
Analysis of responses to a specific usability questionnaire | 3 months
  Eight questions for each connected device and the smartphone application : Level of difficulty in using the connected devices and application? Level of clarity of instructions for use of these connected devices? How much benefit is there from using this type of connected device? Would the patient be willing to pay € 50 or € 100 to keep the device after the study? Does the patient feel confident using connected devices? Has the association of these devices connected to CPAP been proven beneficial? Does the patient think it is necessary to associate connected devices in the management of OSAS? Does the functionality of 3 connected objects and the Sefam Access smartphone application meet the patient's requirements?
Epworth sleepiness scale (ESS) | baseline and 3 months
  The ESS is a self-administered questionnaire with 8 questions. Patients are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 sub-item scores( 0-3) can range from 0 to 24. The higher the ESS score the greater the likelihood that the person has daytime sleepiness. The questionnaire takes no more than 2 or 3 minutes to answer.
Pichot fatigue scale (PWS) | baseline and 3 months
  This is a self-administered questionnaire with 8 questions. Patients are asked to rate, on a 5-point scale (0-4), any habitual feeling of tiredness or weakness while engaged in eight different activities. The Pichot score (the sum of the 8 item sub-scores (0-4) can range from 0 to 32.The higher the score, the more likely that the person suffers from fatigue/ chronic tiredness. The questionnaire takes no more than 2 or 3 minutes to answer.
Assessment of health-related quality of life using the EQ-5D questionnaire | baseline and 3 months
  This questionnaire covers five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The scores for these five dimensions can be presented as a health profile or can be converted to a single summary index number
Analysis of all primary and secondary outcome measures at 1 year | 1 year
  At the end of the first 3 months of the study, the connected devices will be left for the patients who will be encouraged to continue using them.
  Reminders will be sent via the via Sefam Access application at 6, 9 and 12 months to encourage the patient to weigh themselves self, measure their blood pressure and to wear their Actimeter (activity monitor)for 1 week.
Predictive factors of CPAP adherence at three-months | 3 months
  Compliance data on CPAP use will be automatically collected by CPAP telemonitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis JLP Pépin, PhD, Principal Investigator — University Hospital, Grenoble; Dany DJ Jaffuel, MD, Principal Investigator — University Hospital, Montpellier; Thibaut TG Gentina, MD, Principal Investigator — Clinique de la Louvière SELARL SPIRAL, Lille; Frédéric FG Gagnadoux, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France

REFERENCES:
- [Background] Levy P, Kohler M, McNicholas WT, Barbe F, McEvoy RD, Somers VK, Lavie L, Pepin JL. Obstructive sleep apnoea syndrome. Nat Rev Dis Primers. 2015 Jun 25;1:15015. doi: 10.1038/nrdp.2015.15. PMID 27188535
- [Background] Malhotra A, Orr JE, Owens RL. On the cutting edge of obstructive sleep apnoea: where next? Lancet Respir Med. 2015 May;3(5):397-403. doi: 10.1016/S2213-2600(15)00051-X. Epub 2015 Apr 14. PMID 25887980
- [Background] Arnaud C, Dematteis M, Pepin JL, Baguet JP, Levy P. Obstructive sleep apnea, immuno-inflammation, and atherosclerosis. Semin Immunopathol. 2009 Jun;31(1):113-25. doi: 10.1007/s00281-009-0148-5. Epub 2009 Apr 29. PMID 19404644
- [Background] Aron-Wisnewsky J, Clement K, Pepin JL. Nonalcoholic fatty liver disease and obstructive sleep apnea. Metabolism. 2016 Aug;65(8):1124-35. doi: 10.1016/j.metabol.2016.05.004. Epub 2016 May 13. PMID 27324067
- [Background] McEvoy RD, Antic NA, Heeley E, Luo Y, Ou Q, Zhang X, Mediano O, Chen R, Drager LF, Liu Z, Chen G, Du B, McArdle N, Mukherjee S, Tripathi M, Billot L, Li Q, Lorenzi-Filho G, Barbe F, Redline S, Wang J, Arima H, Neal B, White DP, Grunstein RR, Zhong N, Anderson CS; SAVE Investigators and Coordinators. CPAP for Prevention of Cardiovascular Events in Obstructive Sleep Apnea. N Engl J Med. 2016 Sep 8;375(10):919-31. doi: 10.1056/NEJMoa1606599. Epub 2016 Aug 28. PMID 27571048
- [Background] Jullian-Desayes I, Joyeux-Faure M, Tamisier R, Launois S, Borel AL, Levy P, Pepin JL. Impact of obstructive sleep apnea treatment by continuous positive airway pressure on cardiometabolic biomarkers: a systematic review from sham CPAP randomized controlled trials. Sleep Med Rev. 2015 Jun;21:23-38. doi: 10.1016/j.smrv.2014.07.004. Epub 2014 Jul 31. PMID 25220580
- [Background] Craig SE, Kohler M, Nicoll D, Bratton DJ, Nunn A, Davies R, Stradling J. Continuous positive airway pressure improves sleepiness but not calculated vascular risk in patients with minimally symptomatic obstructive sleep apnoea: the MOSAIC randomised controlled trial. Thorax. 2012 Dec;67(12):1090-6. doi: 10.1136/thoraxjnl-2012-202178. Epub 2012 Oct 30. PMID 23111478
- [Background] Pepin JL, Tamisier R, Barone-Rochette G, Launois SH, Levy P, Baguet JP. Comparison of continuous positive airway pressure and valsartan in hypertensive patients with sleep apnea. Am J Respir Crit Care Med. 2010 Oct 1;182(7):954-60. doi: 10.1164/rccm.200912-1803OC. Epub 2010 Jun 3. PMID 20522795
- [Background] Chirinos JA, Gurubhagavatula I, Teff K, Rader DJ, Wadden TA, Townsend R, Foster GD, Maislin G, Saif H, Broderick P, Chittams J, Hanlon AL, Pack AI. CPAP, weight loss, or both for obstructive sleep apnea. N Engl J Med. 2014 Jun 12;370(24):2265-75. doi: 10.1056/NEJMoa1306187. PMID 24918371
- [Background] Schwab RJ, Badr SM, Epstein LJ, Gay PC, Gozal D, Kohler M, Levy P, Malhotra A, Phillips BA, Rosen IM, Strohl KP, Strollo PJ, Weaver EM, Weaver TE; ATS Subcommittee on CPAP Adherence Tracking Systems. An official American Thoracic Society statement: continuous positive airway pressure adherence tracking systems. The optimal monitoring strategies and outcome measures in adults. Am J Respir Crit Care Med. 2013 Sep 1;188(5):613-20. doi: 10.1164/rccm.201307-1282ST. PMID 23992588
- [Background] Redline S, Dean D 3rd, Sanders MH. Entering the era of "big data": getting our metrics right. Sleep. 2013 Apr 1;36(4):465-9. doi: 10.5665/sleep.2524. No abstract available. PMID 23564993
- [Background] Hwang D. Monitoring Progress and Adherence with Positive Airway Pressure Therapy for Obstructive Sleep Apnea: The Roles of Telemedicine and Mobile Health Applications. Sleep Med Clin. 2016 Jun;11(2):161-71. doi: 10.1016/j.jsmc.2016.01.008. Epub 2016 Mar 26. PMID 27236054
- [Derived] Coiffier O, Bailly S, Joyeux-Faure M, Tamisier R, Amrani K, Cornu JC, Gentina T, Terrail R, Causse C, Lombardi C, Pengo MF, Parati G, Pepin JL. Home Blood Pressure Trajectories During 6 Months of Continuous Positive Airway Pressure Therapy: Results from the eMEUSE-SANTE and SLEEPCONNECT Clinic. Ann Am Thorac Soc. 2025 Sep 23. doi: 10.1513/AnnalsATS.202505-504OC. Online ahead of print. PMID 40986800